CLINICAL TRIAL: NCT04739631
Title: Efficacy of Acupuncture on Chemotherapy-Induced Peripheral Neuropathy (CIPN): A Phase III, Randomized, Sham-controlled Clinical Trial
Brief Title: Efficacy of Acupuncture on Chemotherapy-Induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-09-005C
Record Dates: First submitted 2021-01-08; First posted 2021-02-04 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Keywords: acupuncture; chemotherapy-induced peripheral neuropathy; neuropathic pain; von-Frey monofilament test; taxane; platinum
MeSH Terms: conditions — Neuralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture group (Experimental): The acupuncture group and the sham-controlled group will receive three therapeutic sessions each week for four weeks, and another two sessions each week for four weeks (a total of 20 sessions at eight weeks). Each group will be followed-up for four weeks, to evaluate the persistent efficacy of acupuncture.The needle set for the sham acupuncture group and the real acupuncture group will use the CASOON Acupuncture Needle (Wuxi Jiajian Medical Instrument Company, limited), which needle size is 0.3 mm×30 mm. The depth of needling varied based on the patient's body sizes. After insertion, the needles were manually manipulated to obtain the De Qi sensation, which was defined as the acupuncturist feeling a tugging or grasping sensation from the needle manipulation and the patient feeling soreness, fullness, heaviness, or local distension at local needling sites.
  Interventions: Other: acupuncture
- sham-controlled group (Placebo Comparator): The sham acupuncture group will be performed by superficial needling with less than 4mm depth. The needling location is about 0.5 cm away from the acupoints. Both the real acupuncture group and the sham acupuncture group received the same treatment protocol.
  Interventions: Other: minimal acupuncture
- waitlist-control group (No Intervention): As an waitlist-control group, no acupuncture will be performed.

INTERVENTIONS:
Other: acupuncture — use disposable sterile needles to insert to the acupuncture point
  Arms: acupuncture group
Other: minimal acupuncture — The sham-controlled group will be performed with minimal acupuncture(superficial needling) at non- acupoints.
  Arms: sham-controlled group

SUMMARY:
The purpose of this study is to assess the neurological efficacy of acupuncture in patients with cancer who experienced peripheral neuropathy, which is induced by chemotherapy.

DETAILED DESCRIPTION:
Background: Chemotherapy may lead to peripheral neuropathy up to 40% in cancer survivors, especially in some types of patients with cancer. The effect of acupuncture, an ancient Chinese medicine technique, was recognized by the World Health Organization (WHO) in the treatment of several diseases. The postulated mechanisms associated with acupuncture in analgesia or neurogenesis are still under investigation. Considering a moderate recommendation for duloxetine in the treatment of chemotherapy-induced peripheral neuropathy (CIPN) based on based on neuropathic pain, and a few treatment options with evidence for CIPN, acupuncture might be another option. Nowadays, only small scale pilot studies provided initial proof of acupuncture in CIPN, particularly in decreasing neuropathic pain and improving neurotoxicity, the study aims to determine the beneficial effects of acupuncture on CIPN with a large-scale, multicenter, randomized sham-controlled clinical trial. Furthermore, the aim of the study will provide evidence for the clinical therapeutic guideline of CIPN in the future.

ELIGIBILITY:
Inclusion criteria:

The study will enroll patients with a symptom of peripheral neuropathy, including paresthesia, numbness, glove-and-stocking sensory loss distribution or pain in four limbs, and meet the following inclusion criteria:

1. All adult cancer patients (Age≧20-year-old) who received chemotherapy regimens, including adjuvant and neoadjuvant therapy
2. Stage I-III cancer patients
3. Completed chemotherapy regimens more than3 months, including Taxanes (paclitaxel or docetaxel), platinum (cisplatin, oxaliplatin, carboplatin)
4. Baseline von Frey Monofilament test (Target force at hand) ≧ 0.07gms
5. Baseline von Frey Monofilament test (Target force at foot) ≧ 0.4gms
6. Eastern Cooperative Oncology Group (ECOG) performance status ≦3
7. Grading of peripheral sensory neuropathy in National Cancer Institute- common terminology criteria for adverse events,v5.0 (NCI-CTCAE5) ≧1
8. Patients were restricted acupuncture treatment for one month before recruitment
9. Written patient informed consent

Exclusion criteria:

Participants with any of the following conditions will be excluded:

1. Uncontrolled Diabetic Mellitus, HbA1c≧7% is inappropriate[19].
2. Diabetic neuropathy diagnosed before receiving chemotherapy
3. Neuropathy from any type of nerve compression (e.g., carpal/tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy)
4. Concomitant with duloxetine, or another analgesia, including Pregabalin, Venlafaxine, Minocycline, Topical gel, Oxycodone, Naloxone, Cannabinoids, and Angiotensin II type 2 receptor antagonist
5. Severe hemorrhagic coagulopathy or bleeding tendency
6. Unstable cardiovascular disease
7. Severe skin lesions around the treatment sites The researchers will exclude any participants considered to be inappropriate for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
FACT-Neurotoxicity subscale(NtxS) | It will be assessed before the first intervention in the first week, after the 12th intervention in the 4th week , after the 20th intervention in the 8th week, and the follow-up assessment in the end of the 12th week. Each intervention is one day.
  The primary outcome will be the change FACT-Neurotoxicity subscale(NtxS) from baseline to 20 sessions at 8th weeks. The neurotoxicity subscale from the FACT/GOG-NTX-13(version 4) contains 13 items assessing numbness, tingling, and discomfort in the hands or feet, difficulty hearing, tinnitus, joint pain or muscle cramps, weakness, or trouble walking, buttoning buttons, or feeling small shapes when placed in the hand. Items are scored from 0-4 (0 = not at all; 4 = very much) and summed (total score range = 0-52). Since no published data are defining a cut-point for determining a clinically important change in the FACT/GOG Ntx score, we defined a 4 point change as a clinically meaningful improvement in patient-reported CIPN-related neurotoxicity outcome . The authorized translated traditional Chinese version will be purchased in this study.

SECONDARY OUTCOMES:
The change of BPI-SF | It will be assessed before the first intervention in the first week, after the 12th intervention in the 4th week , after the 20th intervention in the 8th week, and the follow-up assessment in the end of the 12th week. Each intervention is one day.
  Our secondary outcome will be the change of average pain severity in BPI-SF from baseline to 20 sessions at 8th weeks. BPI-SF is an instrument used to evaluate the severity of pain, including neuropathic pain and the interference on the patients' daily functioning. Items are scored from 0 to 10 (0= no pain; 10= pain as bad as you can imagine). Since not all the patients feel pain in their daily life, we selected the participants who have average pain severity more than 4 points at baseline assessment into the final analysis. The authorized translated traditional Chinese version will be purchased in this study.
The quantitative sensation of touch detection | It will be assessed before the first intervention in the first week, after the 20th intervention in the 8th week, and the follow-up assessment in the end of the 12th week. Each intervention is one day.
  The quantitative sensation of touch detection was used to test sensory levels and obtain objective data on the status of diminishing or returning sensibility. Touch detection was measured using von Frey monofilaments (Semmes-Weinstein Von Frey Aesthesiometer, Stoelting Co. 620 Wheat Lane, Wood Dale, IL, USA), with weights from 0.008 g to 300 g at 8 points. The measuring sites including the bases of the sole, tips of the big toe, palmar sides of hands, and the fingertips of the middle finger. The well-known up-down method applied to measure touch-detection thresholds.
  It will be assessed before the first intervention in the first week, after the 20th intervention in the 8th week, and the follow-up assessment in the end of the 12th week. Each intervention is one day. Each von-Frey test or questionnaire will be performed within seven days from each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No